CLINICAL TRIAL: NCT00362011
Title: Effect of Chia Seeds (Salvia Hispanica L.) on Glucose Control in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 01-062
Record Dates: First submitted 2006-08-08; First posted 2006-08-09 (Estimated); Last update posted 2006-08-09 (Estimated); Status verified 2001-02

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

INTERVENTIONS:
Behavioral: Salba diet

SUMMARY:
The purpose of this study is to determine whether the addition of Salvia hispanica L. Alba (Salba) to the conventional treatment for diabetes is associated with improvement in major and emerging cardiovascular risk factors in people with type 2 diabetes.

DETAILED DESCRIPTION:
Cohort studies have linked consumption of whole grain with a reduction in the risk of developing diabetes and heart disease. Grain of the plant Salvia hispanica alba (Salba) contain a high concentration of ω-3 fatty acids in addition to being a rich source of vegetable protein, fiber, calcium and antioxidants which have cardiovascular protective effect. To address the paucity of randomized, well-controlled clinical studies supporting the long-term cardioprotective benefits of whole grain we investigated the effects of a novel grain Salba in type 2 diabetes.

Comparison(s): Participants on a conventional diabetes diet (50% carbohydrate, 20% protein, 30% fat) receive either addition of Salba or matched control supplement for 12 weeks separated by a 4-week washout period.

ELIGIBILITY:
Inclusion Criteria:

* All men or postmenopausal women with Type 2 diabetes optimally or suboptimally controlled (HbA1C < 9.0%) on oral hypoglycemic agents or diet only were asked to participate.

Exclusion Criteria:

* Those receiving insulin, alpha-glucosidase inhibitors, or hormone replacement therapy, with BMI>38 kg/m2, smoking or significant alcohol intake (>2 drinks/day), serum TG >4.0 mmol/L, and those with complications of diabetes were excluded. Subjects were also excluded if they regularly took fish oil and flax seed supplements or used steroids. Subjects were excluded during the course of the study if there were any changes to their regular antihypertensive, lipid, or oral hypoglycemic medications, if unable to consume >50% of supplements provided, had a significant weight change (defined as >2.5 kg), or if their level of physical activity did not remain constant over the course of the study.

Ages: 35 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2001-03

PRIMARY OUTCOMES:
Hemoglobin A1c

SECONDARY OUTCOMES:
Efficacy - major and emerging risk factors for cardiovascular disease (blood pressure, Hs-C-reactive protein, coagulation factors)
safety (liver, kidney and haemostatic function)
compliance (plasma fatty-acids, returned supplements, diet records, body weight).

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Vuksan, PhD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Vuksan V, Whitham D, Sievenpiper JL, Jenkins AL, Rogovik AL, Bazinet RP, Vidgen E, Hanna A. Supplementation of conventional therapy with the novel grain Salba (Salvia hispanica L.) improves major and emerging cardiovascular risk factors in type 2 diabetes: results of a randomized controlled trial. Diabetes Care. 2007 Nov;30(11):2804-10. doi: 10.2337/dc07-1144. Epub 2007 Aug 8. PMID 17686832